CLINICAL TRIAL: NCT00390325
Title: Phase II Study of Sorafenib (BAY 43-9006) in Patients With Metastatic Medullary Thyroid Carcinoma
Brief Title: Sorafenib Tosylate in Treating Patients With Metastatic, Locally Advanced, or Recurrent Medullary Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00196; NCI-2009-00196 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006C0050; NCI-7609; CDR0000507441; OSU 06054 / IRB 2006C0050; 7609 (Other: Ohio State University Comprehensive Cancer Center); 7609 (Other: CTEP); N01CM00070 (NIH); N01CM62207 (NIH); P30CA016058 (NIH); NCT01645631 (obsolete NCT alias)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Hereditary Thyroid Gland Medullary Carcinoma; Locally Advanced Thyroid Gland Medullary Carcinoma; Multiple Endocrine Neoplasia Type 2A; Multiple Endocrine Neoplasia Type 2B; Recurrent Thyroid Gland Medullary Carcinoma; Sporadic Thyroid Gland Medullary Carcinoma; Stage III Thyroid Gland Medullary Carcinoma AJCC v7; Stage IV Thyroid Gland Medullary Carcinoma AJCC v7; Stage IVA Thyroid Gland Medullary Carcinoma AJCC v7; Stage IVB Thyroid Gland Medullary Carcinoma AJCC v7; Stage IVC Thyroid Gland Medullary Carcinoma AJCC v7
MeSH Terms: conditions — Familial medullary thyroid carcinoma; Multiple Endocrine Neoplasia Type 2a; Multiple Endocrine Neoplasia Type 2b; Carcinoma, Medullary | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive sorafenib tosylate PO BID in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sorafenib Tosylate

INTERVENTIONS:
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This phase II trial studies how well sorafenib tosylate works in treating patients with medullary thyroid cancer that has spread to other parts of the body (metastatic), spread to the tissue surrounding the thyroid (locally advanced), or has returned after a period of improvement (recurrent). Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess objective response rate of sorafenib tosylate (sorafenib [BAY 43-9006]) in metastatic medullary thyroid carcinoma in setting of inherited tumor syndromes, such as multiple endocrine neoplasia (MEN) 2A, MEN 2B, or familial medullary thyroid carcinoma (FMTC).

II. To assess objective response rate of sorafenib (BAY 43-9006) in sporadic metastatic medullary thyroid carcinoma.

SECONDARY OBJECTIVES:

I. To assess toxicity of sorafenib (BAY 43-9006) in patients with metastatic medullary thyroid carcinoma.

II. Measure serum tumor markers calcitonin and carcinoembryonic antigen (CEA) pre-, during, and post-treatment to correlate with disease response.

III. Correlate nuclear medicine functional imaging (fludeoxyglucose F 18 [F-18 fluorodeoxyglucose] positron emission tomography [PET] scan) data obtained at pre-, during, and post-treatment with tumor response.

IV. Correlate dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) data obtained at pre-, during, and post-treatment with changes in tumor permeability and vascularity with tumor response.

V. Perform pharmacogenomic studies on procured peripheral blood mononuclear cells (PBMCs) if clinical responses are observed.

VI. To correlate between the degree of retrovirus-associated sequence (Ras)-mitogen-activated protein kinase (MAPK) signaling inhibition and vascular endothelial growth factor (VEGF) expression in the tumor and clinical response.

VII. To correlate between the presence and type of ret proto-oncogene (RET) gene defects in tumor and clinical response.

OUTLINE:

Patients receive sorafenib tosylate orally (PO) twice daily (BID) in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA SPECIFIC FOR ARM A
* Histologically confirmed medullary thyroid carcinoma under the clinical setting of inherited tumor syndromes, such as multiple endocrine neoplasia (MEN) 2A, MEN 2B, or familial medullary thyroid carcinoma (FMTC)
* ELIGIBILITY CRITERIA SPECIFIC FOR ARM B
* Histologically confirmed medullary thyroid carcinoma under the clinical setting of sporadic medullary thyroid carcinoma (MTC)
* ELIGIBILITY CRITERIA COMMON FOR ARMS A AND B
* Patients must have measurable disease
* Metastatic and/or locally advanced or locally recurrent disease
* Oral or intravenous (IV) bisphosphonates therapy will be allowed for patients with bony metastasis at the investigator's discretion; bisphosphonate usage should be recorded if used since these agents may have anti-farnesyl transferase activity and may have some therapeutic effect in combination with sorafenib
* Life expectancy must be >= six months
* Patients must have an Eastern Cooperative Oncology Group performance status 0-2
* Leukocytes >= 2,000/uL (10 days prior to patient enrollment)
* Absolute neutrophil count >= 1,000/uL (10 days prior to patient enrollment)
* Platelets >= 100,000/uL (10 days prior to patient enrollment)
* Total bilirubin =< within 2 x upper limit of normal (10 days prior to patient enrollment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< within 3 x upper limit of normal (10 days prior to patient enrollment)
* Serum creatinine within normal institutional limits OR creatinine clearance > 30 mL/min (by Cockcroft-Gault formula) (10 days prior to patient enrollment)
* The effects of sorafenib (BAY 43-9006) on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because kinase inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 30 days after completion of therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* EXCLUSION CRITERIA FOR ARM A AND B
* Patients who have had systemic anti-tumor therapy (such as chemotherapy, biologic modifiers or antiangiogenic therapy) within 4 weeks (6 weeks if nitrosourea or mitomycin chemotherapy) prior to study entry
* Patients who have had external beam radiation therapy within 1 week or if the adverse events associated with radiation are not resolved to grade 1 or less prior to study entry
* Prior therapy with sorafenib (BAY 43-9006), ZD 6474 or AMG-706
* Patients currently receiving any other tumor-specific therapy for thyroid cancer or investigational therapy; patients receiving adjuvant hormonal therapy for a second primary (such as breast cancer or prostate cancer) are allowed to participate as far as there are no known drug interactions
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib (BAY 43-9006)
* Patients unable to swallow sorafenib tablets (e.g. any condition that impairs patient's ability to swallow pills)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with any evidence of a bleeding diathesis
* Patients actively receiving anticoagulation with therapeutic intent; prophylactic anticoagulation (i.e. low dose warfarin) or venous or arterial access devices is allowed provided that the prothrombin time (PT), international normalized ratio (INR) or partial thromboplastin time (PTT) are normal
* Pregnant women or women who are breast-feeding are excluded from this study because sorafenib (BAY 43-9006) is an investigational agent and teratogenicity has not been evaluated yet; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sorafenib (BAY 43-9006), breastfeeding should be discontinued if the mother is treated with sorafenib (BAY 43-9006)
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy because of possible pharmacokinetic interactions with sorafenib (BAY 43-9006); patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Patients taking the cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine, or phenobarbital), rifampin or St. John's wort due to potential drug interactions with sorafenib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-11-03 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavana Konda, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 2006 and January 2008
Groups:
- Arm A (Hereditary MTC); Arm B (Sporadic MTC): Sorafenib (BAY 43-9006) was administered at the dose of 400 mg orally twice a day on a continuous basis.
Period: Overall Study
Arm/Group | Arm A (Hereditary MTC) | Arm B (Sporadic MTC)
Started | 5 | 16
Completed | 5 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Hereditary MTC) | Arm B (Sporadic MTC) | Total
Number analyzed (Participants) | 5 | 16 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 8
  >=65 years | 3 | 10 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 11 | 11
  Male | 5 | 5 | 10
Race/Ethnicity, Customized [Number; unit: patients]
  White | 5 | 13 | 18
  Nonwhite | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 16 | 21

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate of Sorafenib Tosylate in Metastatic Medullary Thyroid Carcinoma in Setting of Inherited Tumor Syndromes as Well as in Setting of Sporadic Medullary Thyroid Cancer
Description: Measured using MRI scans. Determined using Response Evaluation Criteria in Solid Tumors/World Health Organization response criteria. 95% confidence interval will be calculated to estimate the frequency of response.
Time Frame: Up to 4 weeks after last dose of sorafenib tosylate
Population: 1 patient was not evaluable for RECIST evaluation in Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Hereditary MTC) | Arm B (Sporadic MTC)
Number analyzed (Participants) | 5 | 15
Participants | 1 | 1

2. Secondary Outcome: Number of Patients With Decreased Calcitonin Levels
Description: Identifying the number of patients with decreased calcitonin levels
Time Frame: Up to 4 weeks after last dose of sorafenib tosylate
Population: 1 patient was not evaluable in Arm B
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Hereditary MTC): Arm A:
  Sorafenib (BAY 43-9006) was administered at the dose of 400 mg orally twice a day on a continuous basis.
- Arm B (Sporadic MTC): Arm B:
  Sorafenib (BAY 43-9006) was administered at the dose of 400 mg orally twice a day on a continuous basis.
Arm/Group | Arm A (Hereditary MTC) | Arm B (Sporadic MTC)
Number analyzed (Participants) | 5 | 15
Participants | 5 | 11

3. Secondary Outcome: Patient With Decreased Carcinoembryonic Antigen (CEA) Levels
Description: Identify the number of patients with decreased Carcinoembryonic Antigen (CEA) levels
Time Frame: Up to 4 weeks after last dose of sorafenib tosylate
Population: 1 patient was not evaluable in Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Hereditary MTC) | Arm B (Sporadic MTC)
Number analyzed (Participants) | 5 | 15
Participants | 4 | 8

4. Secondary Outcome: Percent of Baseline Dynamic-Contrast Enhanced Magnetic Resonance Imaging (DCE-MRI) Exchange Rate Constant (Kep)
Description: Median decrease in exchange rate Kep in index lesions
Time Frame: Up to 4 weeks after last dose of sorafenib tosylate
Population: kep [exchange rate constant]
Measure: Median (Full Range); unit: percentage change
Groups:
- Arm A (Hereditary MTC) and Arm B (Sporadic MTC): Arm A:
  Sorafenib (BAY 43-9006) was administered at the dose of 400 mg orally twice a day on a continuous basis.
  Arm B:
  Sorafenib (BAY 43-9006) was administered at the dose of 400 mg orally twice a day on a continuous basis.
Arm/Group | Arm A (Hereditary MTC) and Arm B (Sporadic MTC)
Number analyzed (Participants) | 10
percentage change | 79 [25 to 96]

5. Secondary Outcome: Degree of Ras-MAPK Signaling Inhibition in the Tumor
Description: Identify the number of patients with degree of Ras-MAPK signaling inhibition
Time Frame: Up to 4 weeks after last dose of sorafenib tosylate
Population: Due to low tumor cellularity in the samples obtained, such evaluation was not possible
Arm/Group | Arm A (Hereditary MTC) | Arm B (Sporadic MTC)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Degree of Vascular Endothelial Growth Factor (VEGF) Expression in the Tumor
Description: Correlated with clinical response.
Time Frame: Up to 4 weeks after last dose of sorafenib tosylate
Population: No data available
Groups:
- Arm A: MTC in setting of inherited syndromes (MEN-2A, 2B or FMTC) plus Measurable disease Plus No prior ZD6474 or AMG 706
- Arm B: MTC in setting of sporadic ds plus Measurable disease Plus No prior ZD6474 or AMG 706
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Standardized Uptake Value (SUV Max) as Measured by Fludeoxyglucose F-18 Positron Emission Tomography (PET)
Description: Identify the median SUV at baseline and 8 week follow up as measured by Fludeoxyglucose F-18 Positron Emission Tomography (PET).
Time Frame: Up to 4 weeks after last dose of sorafenib tosylate
Measure: Median (Full Range); unit: maximum SUV
Arm/Group | Arm A (Hereditary MTC) and Arm B (Sporadic MTC)
Number analyzed (Participants) | 9
maximum SUV
  Baseline | 3.73 [2.84 to 4.63]
  8 week follow up | 2.94 [2.24 to 3.88]

8. Secondary Outcome: Number of Patients With Toxicity, Graded Using the Revised National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0
Description: Toxicities were graded for patients using the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Time Frame: Up to 4 weeks after last dose of sorafenib tosylate
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Hereditary MTC) and Arm B (Sporadic MTC)
Number analyzed (Participants) | 21
Participants
  Diarrhea | 10
  Oral cavity pain | 13
  Alopecia | 16
  Hypertension | 10
  HFSR | 14
  Pulmonary Embolism | 5

9. Secondary Outcome: Number of Participants With Ret Proto-Oncogene (RET) Gene Defects in the Tumor
Description: Percent of patients with RET mutations
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Hereditary MTC) | Arm B (Sporadic MTC)
Number analyzed (Participants) | 5 | 12
Participants | 5 | 10

10. Secondary Outcome: Selected Polymorphisms of Genes Influencing Sorafenib Tosylate Metabolism and/or Resistance Genes That May Predict Response or Toxicity
Description: Changes will be correlated with toxicity and clinical response to therapy.
Time Frame: Baseline
Population: Due to low tumor cellularity in the samples obtained, such evaluation was not possible
Arm/Group | Arm A (Hereditary MTC) | Arm B (Sporadic MTC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All patients will be evaluable for toxicity from the time of their first treatment with sorafenib (BAY 43-9006) until off study, up to 4 weeks after last dose of sorafenib tosylate", "through study completion, an average of 1 year.
Description: The National Cancer Institutes Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 was utilized for adverse event reporting
Arm/Group | Arm A (Hereditary MTC) and Arm B (Sporadic MTC)
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Hereditary MTC) and Arm B (Sporadic MTC) (N=21)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Perforation, GI-small bowel (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — Infection with normal ANC or Grade 1 or 2 neutrophils-Colon
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Thrombosis/Thrombus/embois (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Hereditary MTC) and Arm B (Sporadic MTC) (N=21)
Weight loss (General disorders) | 10 (10)
Anorexia (Gastrointestinal disorders) | 8 (8)
Fatigue (General disorders) | 7 (7)
Taste Changes (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 17 (17)
Oral Cavity Pain (Gastrointestinal disorders) | 13 (13)
Mucositis (Gastrointestinal disorders) | 10 (10)
Flatulence (Gastrointestinal disorders) | 8 (8)
Abdominal pain or cramping (Gastrointestinal disorders) | 6 (6)
Abdominal bloating (Gastrointestinal disorders) | 4 (4)
Nausea (General disorders) | 3 (3)
Heartburn (Gastrointestinal disorders) | 2 (2)
HFSR (Skin and subcutaneous tissue disorders) | 19 (19) — hand-foot-skin reaction
Alopecia (Skin and subcutaneous tissue disorders) | 16 (16)
Rash (Skin and subcutaneous tissue disorders) | 14 (14)
Nail Changes (Skin and subcutaneous tissue disorders) | 10 (10)
Dry skin/scalp (Skin and subcutaneous tissue disorders) | 10 (10)
Skin lesions/sores (Skin and subcutaneous tissue disorders) | 8 (8) — non HFSR
Scalp pruritis (Skin and subcutaneous tissue disorders) | 7 (7)
Photosensitivity (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 11 (11)
Flushing (Vascular disorders) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Muscle pain or cramping (Musculoskeletal and connective tissue disorders) | 11 (11)
Joint pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Scalp pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Dizziness (Nervous system disorders) | 3 (3)
Infection (Infections and infestations) | 6 (6)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Leukopenia (Investigations) | 11 (11)
Neutropenia (Investigations) | 7 (7)
Lymphopenia (Investigations) | 3 (3)
Thrombocytopenia (Injury, poisoning and procedural complications) | 11 (11)
Anemia (Blood and lymphatic system disorders) | 8 (8)
AST (Investigations) | 9 (9)
LDH (Investigations) | 13 (13)
ALT (Investigations) | 8 (8)
Bilirubin (Investigations) | 4 (4)
Alkaline phosphatase (Investigations) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (12)
Hyponatremia (Metabolism and nutrition disorders) | 12 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT00390325/Prot_SAP_000.pdf